CLINICAL TRIAL: NCT00818298
Title: 24-Hour Time Course of Striatal Dopamine D2 Receptor Occupancy of Ziprasidone: A PET Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre for Addiction and Mental Health (Other)
Collaborators: Pfizer (Industry)
Responsible Party: Principal Investigator, David Mamo, Psychiatrist, Centre for Addiction and Mental Health
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 245/2008
Record Dates: First submitted 2009-01-06; First posted 2009-01-07 (Estimated); Last update posted 2012-07-09 (Estimated); Status verified 2012-07

CONDITIONS: Schizophrenia; Schizoaffective Disorder
Keywords: schizophrenia; schizoaffective disorder; PET Scan; ziprasidone; dopamine; D2; receptor; antagonist; occupancy; dissociation; affinity; constant; Ki; ligand; raclopride; half-life; striatal; plasma dynamics; central dynamics; plasma drug level; compliance; antipsychotic; pharmacotherapy; twice daily dosing; BID dosing; once daily dosing; od dosing; qd dosing; dosing schedule
MeSH Terms: conditions — Schizophrenia; Psychotic Disorders; Dissociative Disorders; Patient Compliance | interventions — ziprasidone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental): ziprasidone
  Interventions: Drug: ziprazidone

INTERVENTIONS:
Drug: ziprazidone — Up to and including the time of the third PET scan, subjects will be titrated to 60 mg BID of ziprazidone. Thereafter they will receive 20-80 mg BID of ziprazidone, according to clinical effectiveness and side effects.

SUMMARY:
Ziprasidone is recommended to be dosed twice daily for the treatment of schizophrenia, based on peripheral pharmacokinetics and a knowledge of its half life in plasma level (5-10 hours). However, the plasma kinetics do not always mirror what occurs in the brain. Antipsychotics with a high-affinity at D2 receptors attach for a relatively long time to their binding sites even after plasma levels declined. Based on this observation, another antipsychotic with a similar high-affinity at D2 receptors, ziprasidone, would also be expected to keep a sufficiently high D2 receptor occupancy even 24 hours after the last dose.

Given >60% D2 occupancy is required to maximize chance of therapeutic efficacy, it would be valuable to assess the D2 receptor occupancy 24 hours postdose to predict the therapeutic effects of once-daily regimen. In this study, we will measure D2 receptor occupancy 6, 12, and 24 hours after the last dose of ziprasidone in patients with schizophrenia.

The hypotheses are as follows: First, based on the known affinity of ziprasidone, the dopamine D2 occupancy 24 hours after the last administered dose of 80 mg will be >60%. Second, the difference in dopamine D2 occupancy between scan at 6 hours and 24 hours will be less than 15%. Third, the difference in dopamine D2 occupancy between scan at 12 hours and 24 hours will be less than 10%. Fourth, ED50 24 hours post dose will be higher that those 6 and 12 hours postdose.

DETAILED DESCRIPTION:
PET studies have demonstrated a therapeutic window of dopamine D2 receptor occupancy (60-80%) in patients with schizophrenia. This observation has been used to predict the therapeutic dose range. Ziprasidone is recommended to be dosed twice daily, based on a knowledge of its half life in plasma level (5-10 hours). However, the plasma kinetics do not always mirror the central kinetics. Antipsychotics with a high-affinity at D2 receptors like risperidone attach for a relatively long time to their binding sites even after plasma levels declined. Based on this observation, another antipsychotic with a similar high-affinity at D2 receptors, ziprasidone, would also be expected to keep a sufficiently high D2 receptor occupancy even 24 hours after the last dose. Given >60% D2 occupancy is required to maximize chance of therapeutic efficacy, it would be valuable to assess the D2 receptor occupancy 24 hours postdose to predict the therapeutic effects of once-daily regimen.

To date, there is no published report to examine D2 receptor occupancy of ziprasidone 24 hours after the last dose in patients with schizophrenia. This study will provide information on 24-hour time course of D2 occupancy of this drug, with which the dissociation between peripheral and central kinetics of this drug will be discussed. The results of this study will also test the feasibility of once daily dosing of ziprasidone, which will directly serve to guide physicians in clinical practice. Furthermore, the findings of this study will elucidate the relationship between D2 receptor occupancy and long-term outcome.

The primary objective to determine the difference in dopamine D2 occupancy of ziprasidone at expected peak plasma levels (6 hours) and 12 and 24 hours postdose. The secondary objectives are to compare ED50 (the plasma levels of ziprasidone resulting in 50% maximal receptor occupancy) 24 hours postdose with those 6 and 12 hours postdose.

Male or female patients aged 18-60 years suffering from schizophrenia or schizoaffective disorder will be eligible to participate in this study (Visit 1). Following the baseline clinical assessments (Visit 2), previous antipsychotics will be discontinued while initiating ziprasidone at 20mg BID and subsequently increasing the dose to 60mg BID (Visit 2-4). For patients already treated with ziprasidone 60 mg BID, no titration will be necessary. If patients are on a lower dose, they will only be included in the study if the treating clinician recommends an increase of the dose to 60 mg BID. Participants will undergo a total of 3 raclopride PET scans (6, 12, and 24 hours postdose) (Visits 5-7) after they have been on ziprasidone for at least 14 days. Psychopathology and side effects will also be assessed on these PET visits. MRI scan will be completed when possible (Visit 8). In the subsequent 6-month follow-up phase (Visit 9-17), participants will have clinical assessments biweekly in the first 3 months and monthly in the following three months. The dose will be titrated according to clinical response and tolerability in an open-labeled manner to a maximum dose of 80 mg BID.

ELIGIBILITY:
Inclusion Criteria:

* Age of 18 - 60 years.
* DSM-IV/SCID diagnosis of schizophrenia, schizoaffective disorder, schizophreniform disorder, delusional disorder, or psychotic disorder NOS
* In- or outpatients
* Physician-of-record's agreement to switch a previous antipsychotic to ziprasidone due to concern about tolerability/ineffectiveness/potential side effects of the previous drug when prescribed

Exclusion Criteria:

* Incapacity to provide consent to psychiatric treatment
* Participation in this study would result in exceeding the annual radiation dose limits (20 mSv) for human subjects participating in research studies.
* Substance abuse or dependence (within past six months)
* Positive urine drug screen
* Positive serum pregnancy test at screening or positive urine pregnancy test before PET scan
* History of clinically significant physical illness or risk factors for drug-induced arrhythmias secondary to QT/QTc interval prolongation
* Presence of risk factors for significant electrolyte disturbances, including diuretic therapy, protracted diarrhea/vomiting, water intoxication, eating disorder, and alcoholism
* A known history of QT prolongation (including congenital long QT syndrome), recent acute myocardial infarction or uncompensated heart failure
* Clinically significant ECG abnormality at screening including a QT/QTc of 450 msec and greater
* Being treated with dofetilide, sotalol, quinidine, other Class Ia and III anti-arrhythmics, sparfloxacin, gatifloxacin, moxifloxacin, halofantrine, mefloquine, pentamidine, arsenic trioxide, levomethadyl acetate, dolasetron mesylate, probucol, tacrolimus, methadone, or clozapine
* A previous history of intolerance or hypersensitivity to ziprasidone or lactose
* History of treatment with long-acting (depot) neuroleptic antipsychotic medication within 6 months
* Subjects at immediate risk of committing harm to self or others
* Metal implants or a pace-maker that would preclude the MRI scan
* History of head trauma resulting in loss of consciousness > 30 minutes that required medical attention
* Unstable physical illness or significant neurological disorder including a seizure disorder
* Size of head, neck, and body being unable to fit PET and MRI scanners
* Refusal to give consent to investigator to communicate with physician of record for the entire duration of the study
* Psychiatric concerns raised by the physician-of-record regarding participation in the study

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2009-01; Primary Completion 2011-01 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
PET Scan | intermittent

CONTACTS AND LOCATIONS:
Overall Officials: David Mamo, MD, MSc, Principal Investigator — Centre for Addiction and Mental Health
Locations (1):
- Centre for Addiction and Mental Health - PET Centre, Toronto, Ontario, Canada

REFERENCES:
- [Derived] Suzuki T, Graff-Guerrero A, Uchida H, Remington G, Caravaggio F, Borlido C, Pollock B, Mulsant B, Deluca V, Ismail Z, Mamo D. Dopamine D(2)/(3) occupancy of ziprasidone across a day: a within-subject PET study. Psychopharmacology (Berl). 2013 Jul;228(1):43-51. doi: 10.1007/s00213-013-3012-1. Epub 2013 Feb 17. PMID 23417515
- See also: Information about research at the Centre for Addiction and Mental Health, Canada's largest mental health and addiction teaching hospital. It is fully affiliated with the University of Toronto, and is a PAHO/WHO Collaborating Centre — http://www.camh.net/research